CLINICAL TRIAL: NCT06229847
Title: The Association of Mindful Eating With Current Glycemic Control in Patients With Type 2 Diabetes
Brief Title: Mindful Eating and Current Glycemic Control in Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Goztepe Prof Dr Suleyman Yalcın City Hospital (Other)
Responsible Party: Principal Investigator, Ayse N Erbakan, Principal investigator, Goztepe Prof Dr Suleyman Yalcın City Hospital
Other Study IDs: Mindful Eating-DM
Record Dates: First submitted 2024-01-14; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; mindful eating; glycemic control; BMI
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the association of the level of mindful eating with the current glycemic control in patients with type 2 diabetes. The researchers will compare different glycemic control levels with the participants mindfulness while eating. And secondly, the researchers will compare the levels of eating awareness of those with and without obesity.

DETAILED DESCRIPTION:
In type 2 diabetes, life style adaptations, mainly healthy eating, weight loss or control and exercise constitutes the foundation of type 2 diabetes management. In addition to regulating blood sugar levels, lifestyle modifications play a significant role in controlling risk factors such as hypertension and hyperlipidemia, delaying/preventing complications from developing, and even promoting diabetes regression. It is essential not only to focus on healthy food choices in dietary therapy but also to ensure patients achieve weight loss. Another crucial point is maintaining the continuity of these lifestyle changes.

It is reported that it is quite challenging for patients to make lifestyle changes, adapt to the offered treatments, and furthermore, sustain this as a way of life. Adherence to these dietary changes is crucial for long-term success in managing diabetes and achieving weight loss goals.

In a cross-sectional study conducted by Fanning and colleagues with 148 type 2 diabetic patients, it was found that "conscious eating" is associated with better diet adherence. In a review by Dunn et al., the available data strongly support the necessity of "conscious eating" as part of weight management programs. An American Heart Association statement highlights strong evidence that irregular eating patterns can make it difficult to maintain a healthy cardiometabolic profile, and emphasizes that conscious attention to mealtime and frequency can contribute to a healthier lifestyle and better management of cardiometabolic risk factors.

In this study, the aim was to investigate the degree of eating mindfulness of patients with type 2 diabetes, and compare it between patients who had good glycemic control and patients with poorly controlled glycemic.

ELIGIBILITY:
Inclusion Criteria:

* given consent to the study
* having applied to Diabetes Outpatient Clinic for diabetes management
* having diagnosed with type 2 diabetes for at least 6 months
* having the mental competence to answer the questions in the questionnaire

Exclusion Criteria:

* Inconclusive diagnosis of type 2 diabetes
* having not received or not using any treatment for diabetes

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals attending to the diabetes outpatient clinic with type 2 diabetes diagnosis for at least 6 months, and received treatment for diabetes
Sampling Method: Non-Probability Sample
Enrollment: 448 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
mindful eating, its subgroups and diabetes control in patients with type 2 diabetes | baseline
  To investigate the relationship between mindful eating and its subgroups with glycemic control, as evaluated by HbA1c, in individuals diagnosed with type 2 diabetes for at least 6 months.

SECONDARY OUTCOMES:
mindful eating, its subgroups and the presence of obesity in patients with type 2 diabetes | baseline
  To investigate the relationship between mindful eating and its subgroups with obesity, as evaluated by body mass index, in individuals diagnosed with type 2 diabetes for at least 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe N Erbakan, MD, Principal Investigator — Istanbul Medeniyet University Goztepe Prof Dr Suleyman Yalcın City Hospital
Locations (1):
- Istanbul Medeniyet University Goztepe Research and TRaining Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fanning J, Osborn CY, Lagotte AE, Mayberry LS. Relationships between dispositional mindfulness, health behaviors, and hemoglobin A1c among adults with type 2 diabetes. J Behav Med. 2018 Dec;41(6):798-805. doi: 10.1007/s10865-018-9938-3. Epub 2018 May 25. PMID 29802533
- [Background] Dunn C, Haubenreiser M, Johnson M, Nordby K, Aggarwal S, Myer S, Thomas C. Mindfulness Approaches and Weight Loss, Weight Maintenance, and Weight Regain. Curr Obes Rep. 2018 Mar;7(1):37-49. doi: 10.1007/s13679-018-0299-6. PMID 29446036
- [Background] St-Onge MP, Ard J, Baskin ML, Chiuve SE, Johnson HM, Kris-Etherton P, Varady K; American Heart Association Obesity Committee of the Council on Lifestyle and Cardiometabolic Health; Council on Cardiovascular Disease in the Young; Council on Clinical Cardiology; and Stroke Council. Meal Timing and Frequency: Implications for Cardiovascular Disease Prevention: A Scientific Statement From the American Heart Association. Circulation. 2017 Feb 28;135(9):e96-e121. doi: 10.1161/CIR.0000000000000476. Epub 2017 Jan 30. PMID 28137935
- [Background] Mason AE, Saslow L, Moran PJ, Kim S, Wali PK, Abousleiman H, Hartman A, Richler R, Schleicher S, Hartogensis W, Epel ES, Hecht F. Examining the Effects of Mindful Eating Training on Adherence to a Carbohydrate-Restricted Diet in Patients With Type 2 Diabetes (the DELISH Study): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Feb 20;8(2):e11002. doi: 10.2196/11002. PMID 30545813